CLINICAL TRIAL: NCT00279149
Title: Therapeutic Trial Evaluating Efficacy of Telemedicine (TELESTROKE) in the Management of Patient With Acute Stroke Within 3-hour After Their Symptom Onset Who Are Admitted to a Remote Hospital With no Stroke Unit Facility
Brief Title: TRUST-tPA: Therapeutic Trial Evaluating Efficacy of Telemedicine (TELESTROKE) of Patients With Acute Stroke
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Zakia Idir, Department Clinical Research of Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P 030443
Record Dates: First submitted 2006-01-13; First posted 2006-01-19 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2007-02

CONDITIONS: Acute Stroke
Keywords: Telemedicine; TELESTROKE; symptoms of ischemic stroke since less than 3 hours
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- surgery (Experimental): surgery
  Interventions: Procedure: Visio conference system connected to the Tele-stroke network

INTERVENTIONS:
Procedure: Visio conference system connected to the Tele-stroke network — Visio conference system connected to the Tele-stroke network

SUMMARY:
The objective is to evaluate decision making of i.v. tPA treatment in acute stroke within 3 hours of symptom onset either remotely via videoconferencing system (investigational arm) beginning of treatment on-site and then transfer to stroke unit vs. decision after immediate transfer to stroke unit (usual care arm). Ten remote hospitals are connected to the BICHAT stroke unit. All patients will have stroke unit care at BICHAT hospital. Primary end-point is rankin 0-1 at 3 months.

DETAILED DESCRIPTION:
This study is a therapeutic trial, comparing a TELESTROKE decision making as the tested hypothesis to usual care (immediate transfer to stroke unit). Once the ER doctor in one of the 10 remote hospitals will judge his patient eligible for tPA thrombolysis, he will call the BICHAT stroke unit visio-conference system. Then, according to the randomization list, the patient will be allocated to 'standard care arm' which is the EMEA-approved tPA labeling (i.e., transfer the patient immediately to a stroke unit to have tPA thrombolysis if the patient arrives in due time -before 3 hours of stroke onset) or he will be allocated to 'TELESTROKE ARM"(i.e., remote neurological exam to perform NIHSS, assess the exact time of the first stroke symptoms onset and visualization of brain CT-scan by the vascular neurologist; then start the tPA thrombolysis on site if the indication is confirmed by the vascular neurologist, then transfer the patient to the BICHAT stroke unit). The primary outcome will be Rankin 0-1 (i.e., cured) at 3 months; secondary outcome will be death or dependency at 3 months and the frequency of symptomatic intracranial hemorrhage at 10 days. Patients randomized will be systematically transfer to the BICHAT stroke unit, no matter the received or not tPA thrombolysis, and no matter the study arm, according to the intention-to-treat rule.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years
* symptoms of brain infarction since less than 150 minutes
* NIHSS between 4 and 22
* No brain hemorrhage on contrast CT-scan
* Signed consent form by the patient or his relatives

Exclusion Criteria:

* NIHSS above 22 or coma
* current oral anticoagulant or INR > 1.7
* heparin treatment within the preceding 24 hours or prolonged APTT (>40seconds)
* platelets count < 100 000/mm3
* another stroke or brain trauma within 3 months prior admission
* systolic blood pressure > 185 or diastolic blood pressure > 110 at the time od tPA treatment onset
* neurologic deficit is improving
* history of intracranial hemorrhage
* glycemia less than 0.5g/l or upper than 4g/l after treatment by Actrapid
* epileptic seizure at the time of stroke onset
* Gastro-intestinal or urinary hemorrhage
* Recent myocardial infarction within the last 21 days
* Lumbar puncture or arterial blood sampling in a non compressible vessel within the last 7 days
* Hemophilia
* Pregnancy or breast feeding
* Pericarditis within the last 3 months
* Major surgery within the last 15 days
* History of aortic dissection
* Endocarditis with the last 3 months

Brain CT scan exclusion criteria:

* Mass effect ( tumor, VAM, aneurism )
* Decreased density ( ASPECTS score < 8) or mass effect involving more than 1/3 of the territory of the middle cerebral artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2006-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients cured at 3 months (rankin score 0,1) | at 3 months
  Percentage of patients cured at 3 months (rankin score 0,1)

SECONDARY OUTCOMES:
NIHSS, rankin score ( 0,1,2) and Barthel Index at 3 months , | at 3 months
  NIHSS, rankin score ( 0,1,2) and Barthel Index at 3 months ,
percentage of symptomatic intracranial hemorrhage at 8 days | at 8 days
  percentage of symptomatic intracranial hemorrhage at 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Pierre AMARENCO, Pr,MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (9):
- France (9):
  - Hôpital d'Argenteuil, Emergency Unit, Argenteuil
  - Hôpital Avicenne, Emergency Unit, Bobigny
  - Hôpital Ambroise Paré, Emergency Unit, Boulogne
  - Hôpital Beaujon, Emergency Unit, Clichy
  - Hôpital Louis Mourier, Emergency Unit, Colombes
  - Hôpital de Compiègne, Emergency Unit, Compiègne
  - Hôpital de Lagny sur Marne, Emergency Unit, Lagny
  - BICHAT HOSPITAL Departement of Neurology, Paris
  - Hôpital de Provins, Emergency Unit, Provins

REFERENCES:
- [Derived] Mazighi M, Meseguer E, Labreuche J, Miroux P, Le Gall C, Roy P, Tubach F, Amarenco P. TRUST-tPA trial: Telemedicine for remote collaboration with urgentists for stroke-tPA treatment. J Telemed Telecare. 2017 Jan;23(1):174-180. doi: 10.1177/1357633X15615762. Epub 2016 Jul 9. PMID 26656722